CLINICAL TRIAL: NCT02339207
Title: A Randomized, Double-blind, Placebo-controlled, First-in-human, 3 Part Study of Orally Administered AL-335 to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single Ascending Dosing and Food-effect in Healthy Volunteers, and Multiple Ascending Dosing in Subjects With Chronic Hepatitis C Genotype 1 Infection
Brief Title: First in Human Study of AL-335; Single Dose, Food Effect in Healthy Volunteers; Multiple Doses in Chronic Hepatitis C Genotype 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alios Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AL-335-601
Record Dates: First submitted 2014-12-18; First posted 2015-01-15 (Estimated); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — adafosbuvir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo dosed once in human volunteers in increasing dosages or once daily for seven days in patients with chronic Hepatitis C in increasing dosages.
  Interventions: Drug: AL-335 matching placebo
- AL-335 (Experimental): AL-335 dosed once in human volunteers in increasing dosages or once daily for seven days in patients with chronic Hepatitis C in increasing dosages.
  Interventions: Drug: AL-335

INTERVENTIONS:
Drug: AL-335 matching placebo
  Arms: Placebo
Drug: AL-335
  Arms: AL-335

SUMMARY:
This randomized, double-blind, placebo-controlled, 3-part study will assess the safety, tolerability, and pharmacokinetics of orally administered AL-335 in healthy volunteers (HV) and subjects with CHC infection.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided written consent.
* In the investigator's opinion, the subject is able to understand and comply with protocol requirements, instructions, and protocol stated restrictions and is likely to complete the study as planned.
* Subject is in good health as deemed by the investigator, based on the findings of a medical evaluation including medical history, physical examination, laboratory tests, and ECG.
* Male or female, 18-60 years of age for HV and 18-65 years of age for subjects with CHC.
* Body mass index (BMI) 18-32 kg/m2, inclusive, for HV and 18-35 kg/m2, inclusive, for subjects with CHC. The minimum weight is 50 kg in both populations. No more than 25% of patients in any cohort may be enrolled with a BMI ≥ 30 kg/m2.
* A female subject is eligible to participate in this study if she is of non childbearing potential (defined as females with a documented tubal ligation, bilateral oophorectomy, or hysterectomy) or postmenopausal (defined as 12 months of spontaneous amenorrhea and follicle stimulating hormone (FSH) level within the laboratory's reference range for postmenopausal females). A post-menopausal female receiving hormone replacement therapy who is willing to discontinue hormone therapy 28 days before study drug dosing and agrees to remain off hormone replacement therapy for the duration of the study may be eligible for study participation.
* If male, subject is surgically sterile or practicing specific forms of birth control (as outline in Section 6.2.9) until 90 days after the end of the study.

Additional inclusion criteria for subjects with CHC infection:

* Documentation of Genotype 1 HCV infection for greater than 6 months at dosing
* Screening HCV RNA viral load ≥ 105 IU/mL using a sensitive quantitative assay, such as COBAS® Taqman® HCV Test 2.0

Exclusion Criteria:

1. Clinically significant cardiovascular, respiratory, renal, gastrointestinal, hematologic, neurologic, thyroid, or any other medical illness or psychiatric disorder, as determined by the Investigator and/or Sponsor's Medical Monitor.
2. Positive test for HAV IgM, HBsAg, or HIV Ab. In Parts 1 and 2 positive HCV serology is exclusionary.
3. Any condition that, in the opinion of the investigator, would compromise the study's objectives or the well-being of the subject or prevent the subject from meeting the study requirements.
4. Participation in an investigational drug trial or having received an investigational vaccine within 30 days or 5 half lives (whichever is longer) prior to study medication.
5. Clinically significant abnormal ECG findings. Particularly, a history or family history of prolonged QT syndrome (e.g., torsade de pointes) or sudden cardiac death; or a corrected QT interval (QTc) > 450 milliseconds for male subjects and >470 milliseconds for female subjects at the Screening Visit.
6. Clinically significant blood loss or elective blood donation of significant volume (i.e., > 500 mL) within 60 days of first dose of study drug; > 1 unit of plasma within 7 days of first dose of study drug.
7. Abnormal heart rate, respiratory rate, temperature or blood pressure values outside of the normal range (evaluated in a semi-recumbent or recumbent position after 5 minutes of rest). One repeat measurement after an additional 5 minutes of rest is permitted.
8. Evidence of active infection (other than CHC infection in subjects enrolled in Part 3).
9. Unwilling to abstain from alcohol for 48 hours prior to the start of dosing through the study completion visit.
10. History of regular alcohol intake > 7 units per week of alcohol for females and > 14 units per week for males (one unit is defined as 10 g alcohol) within 3 months of screening visit.
11. For healthy subjects (Parts 1-2), history of regular use of tobacco (i.e., ≥10 cigarettes per day) or nicotine-containing products within 3 months of the screening visit. For subjects with CHC infection, history of regular use of tobacco- or nicotine-containing products is allowed.
12. The subject has a positive pre-study drug screen. A minimum list of drugs that will be screened for includes amphetamines, barbiturates, cocaine, opiates, cannabinoids, phencyclidine (PCP) and benzodiazepines. Subjects with CHC may be included if they have a positive result for cannabinoids at screening. However, they must be willing to abstain from cannabinoid use throughout the duration of the study.
13. In Parts 1-2, the use of concomitant medications, including prescription, over the counter medications, or herbal medications within 14 days prior to the first dose of study medication is excluded, unless approved by the Sponsor's Medical Monitor. PRN use of a nonsteroidal anti inflammatory drug (NSAID) is permitted.
14. For subjects in Part 3, the use of prescription and over the counter medications deemed necessary to maintain the health status of the subject are permitted, if approved by the Sponsor's Medical Monitor. PRN NSAID use is permitted. Further guidance for the use of prior medication in subjects with CHC can be found in Section 5.7.
15. Subjects must not have received any drug known to be a strong inducer or inhibitor of CYP450 enzymes within 2 weeks prior to study drug dosing (Appendix C).
16. Exposure to more than four new investigational entities within 12 months prior to the first dosing day.
17. Abnormal biochemistry or hematology laboratory results obtained at screening. Elevated bilirubin in subjects with suspected Gilbert's disease is allowed.

    Additional exclusion criteria for subjects with CHC infection:
18. History of clinical hepatic decompensation, e.g., variceal bleeding, spontaneous bacterial peritonitis, ascites, hepatic encephalopathy or active jaundice
19. Liver biopsy within two years or Fibroscan evaluation within 6 months prior to randomization that demonstrates cirrhosis (Knodell score >3, Metavir score > 3, Ishak score > 4). Fibroscan liver stiffness score > 10.5 kPa.
20. Prior treatment for CHC
21. Serum alanine aminotransferase (ALT) concentration >5 x ULN
22. Alpha Fetoprotein (AFP) is ≥ ULN, unless the absence of a hepatic mass or lesion is demonstrated by ultrasound within the screening period.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2014-12-31 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2016-05-31 (Actual)

PRIMARY OUTCOMES:
Safety Data: Number and frequency of treatment emergent adverse events, physical examination findings, abnormal vital signs, 12 lead ECG and abnormal clinical laboratory results | From screening to Day 8 (SAD/FE) and Day 21 (MAD)
  Tabulation of the number and frequency of treatment emergent adverse events, physical examination findings, abnormal vital signs, 12 lead ECG and abnormal clinical laboratory results (including chemistry, hematology, and urine).

SECONDARY OUTCOMES:
Single Dose PK: Cmax, tmax, t1/2, CL/F and Vz/F (for AL-335 only), AUC0-inf or AUClast | From dosing to Day 8 visit for each SAD/FE cohort
  PK parameters of AL-335, and metabolites following single dose administration: Cmax, tmax, t1/2, CL/F and Vz/F (for AL-335 only), AUC0-inf or AUClast
Multiple Dose PK: Cmax, tmax, t1/2, AUClast and AUC0 tau | From dosing to final study visit (21 days) for each cohort
  • PK parameters of AL-335, ALS-022399, ALS-022227 (and other metabolites if applicable) following repeat dose administration: Cmax, tmax, t1/2, AUClast and AUC0 tau
Hepatitis C viral levels | From screening to final study visit (21 days) for each cohort
  HCV ribonucleic acid (RNA) viral load change from baseline to final study visit in subjects with CHC infection

CONTACTS AND LOCATIONS:
Locations (3):
- Biotrial, Rennes, Brittany Region, France
- Arensia, Research Institute of Clinical Medicine, Tbilisi, Georgia
- Arensia, Republican Clinical Hospital, Chisinau, Moldova

REFERENCES:
- [Derived] McClure MW, Berliba E, Tsertsvadze T, Streinu-Cercel A, Vijgen L, Astruc B, Patat A, Westland C, Chanda S, Zhang Q, Kakuda TN, Vuong J, Khorlin N, Beigelman L, Blatt LM, Fry J. Safety, tolerability, and pharmacokinetics of AL-335 in healthy volunteers and hepatitis C virus-infected subjects. PLoS One. 2018 Oct 16;13(10):e0204974. doi: 10.1371/journal.pone.0204974. eCollection 2018. PMID 30325939